CLINICAL TRIAL: NCT02154581
Title: Case Selection and Treatment Protocol for Immediate Dental Implants in the Esthetic Zone: A Controlled Clinical Trial
Brief Title: Case Selection and Treatment Protocol for Immediate Dental Implants in the Esthetic Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITI 799_2011; HSC20130085H (Other: UTHSCSA IRB)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Jaw, Edentulous, Partially; Acquired Absence of Single Tooth
Keywords: Dental implants; Esthetic score; Immediate implants; Gingival biotype
MeSH Terms: conditions — Jaw, Edentulous, Partially | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type 1 implant and thin biotype (Active Comparator): In this group, immediate implant placement (SLActive implant) is performed in patients with thin tissue biotype. In addition to implant placement bone grafting of the void between the implant and the fresh extraction socket, bone grafting the buccal aspect of the buccal plate (overcontouring) and soft tissue grafting (connective tissue) are performed.
  Interventions: Device: SLActive implant
- Type 1 implant and thick biotype (Active Comparator): In this group, immediate implant placement (SLActive implant) is performed including bone grafting of the void between the implant and the fresh extraction socket.
  Interventions: Device: SLActive implant

INTERVENTIONS:
Device: SLActive implant
  Other Names: Straumann; Dental Implants; Type 1 implant placement

SUMMARY:
In this study a tooth that needs to be extracted will be replaced by an implant (artificial root) placed at the same appointment as the extraction. The investigators want to observe how the gums change shape with healing in two different scenarios:

1. If the soft tissue around your tooth is thin, following extraction and implant placement an extra soft tissue graft (taken from your palate) in the area in order to increase the thickness of your gums after healing.
2. If the soft tissue around your tooth is thick, the implant will be placed without a soft tissue graft.

Previous studies have shown that both methods work and can give good results. In fact the two methods are used routinely but they have never been compared objectively to one another in the same research study.

The main purpose of this study is to evaluate if there is any difference in terms of esthetic outcomes between these two treatment modalities after a crown has been placed on the implant.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is 18 years or older.
2. Ability to understand and provide informed consent before starting the study.
3. Ability and willingness to comply with all study requirements.
4. The patient, if of child-bearing potential, has a negative urine pregnancy test.
5. Adequate oral hygiene to allow for implant therapy consistent with standards of care.
6. Adequate bone volume to accommodate the planned endosseous dental implant placement according to immediate placement protocols utilizing Straumann Bone Level implants RC (Regular Crossfit) 4.1mm or Bone Level Implant NC (Narrow Crossfit) 3.3 mm at 8, 10,12 or 14mm in length.
7. One tooth in the anterior maxilla (first pre-molar to first pre-molar) requiring extraction resulting in a single- tooth gap planned to be restored with a dental implant as determined by the patient's dental provider.
8. The site to be treated is surrounded by two natural teeth.
9. Except the site to be treated, none of the maxillary incisors, canines and first pre-molars display marginal soft tissue recession.
10. Following extraction, intact extraction socket bony walls are present.
11. Primary stability of implant consistent with standards of care is achieved at the time of implant placement.
12. Patient must be able to pay for fees related to the surgical implant placement related to extraction, grafting of the implant site, and half of the cost of the crown at the time of implant placement.

Exclusion Criteria:

1. Patient reports tobacco use within the last five years. Tobacco use for this study is defined as a current smoking habit with moderate or heavy smoking (more than 10 cigarettes per day) or tobacco chewing use.
2. History of alcoholism or drug abuse within the past 5 years.
3. Severe wear with an etiology of bruxism or clenching habits.
4. Patient has significant untreated periodontal disease (grade III or IV), caries, or clinical or radiographic signs of infection within two adjacent tooth positions of implant area.
5. History of HIV infection, Hepatitis B or C.
6. Patients with a history of systemic disease that precludes standard dental implant therapy or alters daily activities to a level consistent with ASA (American Society of Anesthesiologists) III classification (including cardiovascular, hepatic, renal, gastrointestinal, metabolic, neurologic, pulmonary, endocrine, autoimmune, or psychiatric disorders).
7. Presence of local inflammation or mucosal diseases such as lichen planus.
8. Patient history consistent with high risk for subacute bacterial endocarditis.
9. Current hematological disorder or warfarin (or similar) therapy.
10. Patient has a disease that affects bone metabolism, such as, but not limited to, osteoporosis, hyperthyroidism, hyperparathyroidism, congenital connective tissue disorders (e.g., osteogenesis imperfecta), or Paget's disease.
11. Patient is taking medications or having treatments known to have an effect on bone turnover, including: thiazide diuretics, calcitonin, systemic steroids, bisphosphonates, vitamin D (>800 IU/day), estrogen or progesterone therapy.
12. Current steroid treatment: defined as any person who within the last two years has received for two weeks a dose equivalent to 20 mg hydrocortisone.
13. Patient currently undergoing chemotherapy.
14. Patient history of radiation treatment to the head or neck.
15. Physical or mental handicaps that would interfere with patient's ability to exercise good oral hygiene on a regular basis.
16. Use of any investigational drug or device within the 30 day period immediately prior to implant surgery.
17. Patient is pregnant.
18. Extraction sites having anatomic conditions that preclude immediate implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-01; Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Huynh-Ba, DDS, MS, Principal Investigator — UTHSCSA Department of Periodontics
Locations (1):
- Graduate Periodontics, Dental School, UTHSCSA, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started in January 2013 and ended in November 2016. All patient were recruited at the University of Texas Health San Antonio, Department of Periodontics.
Pre-assignment Details: No patient was excluded prior to group assignment.
Groups:
- Type 1 Implant and Thick Biotype: In this group, immediate implant placement (SLActive implant) is performed including bone grafting of the void between the implant and the fresh extraction socket.
  SLActive implant
- Type 1 Implant and Thin Biotype: In this group, immediate implant placement (SLActive implant) is performed in patients with thin tissue biotype. In addition to implant placement bone grafting of the void between the implant and the fresh extraction socket, bone grafting the buccal aspect of the buccal plate (overcontouring) and soft tissue grafting (connective tissue) are performed.
  SLActive implant
Period: Overall Study
Arm/Group | Type 1 Implant and Thick Biotype | Type 1 Implant and Thin Biotype
Started | 21 | 20
Completed | 14 | 12
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 7 | 8

BASELINE CHARACTERISTICS:
Population: Each patient received one dental implant which was included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 1 Implant and Thick Biotype | Type 1 Implant and Thin Biotype | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Customized [Count of Participants; unit: Participants]
  Participants over 18 years of age | 14 | 12 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 6 | 2 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Mid Facial Mucosal Level at Implant Site
Description: Baseline will be at the time of crown delivery. Thereafter, the mid facial mucosal level at implant site will be recorded at 3, 6, 12 months after crown delivery.
Time Frame: Change from Baseline to 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Type 1 Implant and Thick Biotype | Type 1 Implant and Thin Biotype
Number analyzed (Participants) | 14 | 12
mm | 0.36 (1.29) | 0.49 (1.27)

2. Secondary Outcome: PES/WES (Pink Esthetic Score, White Esthetic Score).
Description: Baseline will be at the time of crown delivery. Secondary outcome measures will be recorded at 12 months after crown delivery. The PES (Pink Esthetic Score) and WES (White Esthetic Score) scales are 10 point scales, made up of 5 categories, each with a 2 point value. Each category is scored out of 2, and the scores totaled to give an optimal score out of 10, and then the two scores (PES and WES) added to give a total score out of 20, with 20 being the highest possible score (best outcome) and 0 being the worst outcome.
Time Frame: Approximately 1 year after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Type 1 Implant and Thick Biotype | Type 1 Implant and Thin Biotype
Number analyzed (Participants) | 14 | 12
score on a scale | 12.07 (2.87) | 11.64 (3.22)

3. Secondary Outcome: Probing Depth
Description: Baseline will be at the time of crown delivery. Secondary outcome measures will be recorded at baseline, 3 and 12 months after crown delivery. The measurement of the pocket around the implanted tooth, measured with a graduated probe. A healthy pocket depth is around 3 mm with no bleeding during the measurement process. The values are totaled and a mean score of all the readings is reported.
Time Frame: Up to 1 year after baseline
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Type 1 Implant and Thick Biotype: In this group, immediate implant placement (SLActive implant) is performed in patients with thin tissue biotype. In addition to implant placement bone grafting of the void between the implant and the fresh extraction socket, bone grafting the buccal aspect of the buccal plate (overcontouring) and soft tissue grafting (connective tissue) are performed.
  SLActive implant
- Type 1 Implant and Thin Biotype: In this group, immediate implant placement (SLActive implant) is performed including bone grafting of the void between the implant and the fresh extraction socket.
  SLActive implant
Arm/Group | Type 1 Implant and Thick Biotype | Type 1 Implant and Thin Biotype
Number analyzed (Participants) | 14 | 12
mm
  Baseline at Crown delivery (Mesial measurement) | 3.14 (0.77) | 2.50 (1.24)
  3 months (Mesial) | 3.21 (0.70) | 2.92 (1.16)
  12 months (Mesial) | 3.29 (0.83) | 2.42 (1.31)
  Baseline at Crown Delivery (Distal Measurement) | 3.43 (0.85) | 2.33 (0.49)
  3 months (distal) | 3.43 (1.02) | 2.08 (0.51)
  12 months (distal) | 3.36 (1.01) | 2.42 (0.51)
  Baseline at Crown Delivery (Buccal Measurement) | 2.93 (1.14) | 1.75 (0.75)
  3 months (Buccal) | 3.07 (1.27) | 1.75 (0.75)
  12 months (Buccal) | 3.21 (1.58) | 1.92 (0.79)
  Baseline at Crown Delivery (Proximal measurement) | 2.64 (0.50) | 2.00 (0.85)
  3 months (proximal) | 2.79 (0.80) | 1.67 (0.78)
  12 months (proximal) | 2.21 (0.70) | 1.75 (0.97)

4. Secondary Outcome: Modified Plaque Index
Description: Baseline will be at the time of crown delivery. Secondary outcome measures will be recorded at 3, 6, 12 months after crown delivery. Measurement of amount of plaque build-up on teeth, using a scale of 0 (no plaque detection), to 3 (an abundance of soft matter). The scores are totaled and a mean score reported.
Time Frame: Up to 1 year after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Type 1 Implant and Thick Biotype | Type 1 Implant and Thin Biotype
Number analyzed (Participants) | 12 | 14
score on a scale
  Baseline crown delivery (Mesial measurement) | 0.29 (0.61) | 0.42 (1.00)
  3 months (Mesial) | 0.36 (0.63) | 0.08 (0.29)
  12 months (Mesial) | 0.50 (0.76) | 0.00 (0.00)
  Baseline at Crown Delivery (Distal Measurement) | 0.36 (0.50) | 0.17 (0.58)
  3 months (distal) | 0.29 (0.61) | 0.17 (0.39)
  12 months (distal) | 0.29 (0.61) | 0.08 (0.29)
  Baseline at Crown Delivery (Buccal Measurement) | 0.14 (0.36) | 0.08 (0.29)
  3 months (Buccal) | 0.14 (0.53) | 0.00 (0.00)
  12 months (Buccal) | 0.29 (0.47) | 0.00 (0.00)
  Baseline at Crown Delivery (Proximal measurement) | 0.36 (0.50) | 0.00 (0.00)
  3 months (proximal) | 0.07 (0.27) | 0.00 (0.00)
  12 months (proximal) | 0.21 (0.58) | 0.00 (0.00)

5. Secondary Outcome: Modified Bleeding Index
Description: Baseline will be at the time of crown delivery. Secondary outcome measures will be recorded at 3, 6, 12 months after crown delivery. Bleeding from the gums is measured on probing the gum and measured on scale of 0 to 5, with 0 being the best outcome, with no bleeding, and 5 being the worst outcome, with spontaneous bleeding. The scores are totaled and a mean score reported.
Time Frame: Up to 1 year after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Type 1 Implant and Thick Biotype | Type 1 Implant and Thin Biotype
Number analyzed (Participants) | 14 | 12
units on a scale
  Baseline crown delivery (Mesial measurement) | 0.43 (0.65) | 0.00 (0.00)
  3 months (Mesial) | 0.29 (0.47) | 0.08 (0.29)
  12 months (Mesial) | 0.29 (0.47) | 0.08 (0.29)
  Baseline at Crown Delivery (Distal Measurement) | 0.43 (0.51) | 0.17 (0.39)
  3 months (distal) | 0.14 (0.36) | 0.08 (0.29)
  12 months (distal) | 0.29 (0.47) | 0.17 (0.39)
  Baseline at Crown Delivery (Buccal Measurement) | 0.21 (0.58) | 0.17 (0.39)
  3 months (Buccal) | 0.36 (0.50) | 0.25 (0.62)
  12 months (Buccal) | 0.64 (0.9) | 0.00 (0.00)
  Baseline at Crown Delivery (Proximal measurement) | 0.14 (0.36) | 0.00 (0.00)
  3 months (proximal) | 0.36 (0.50) | 0.00 (0.00)
  12 months (proximal) | 0.29 (0.47) | 0.00 (0.00)

6. Secondary Outcome: Radiographic Bone Level
Description: Baseline will be at the time of crown delivery. Secondary outcome measures will be recorded at baseline 3, and 12 months after crown delivery. Radiographic bone measurements recorded following final restoration placement (baseline), after 3 and 12 months of loading, and change between these time points. A positive value indicates bone loss and a negative value indicates bone gain. BIC (Bone implant contact)= Distance from implant shoulder to first bone to implant contact.
Time Frame: Up to 1 year after baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Type 1 Implant and Thick Biotype | Type 1 Implant and Thin Biotype
Number analyzed (Participants) | 14 | 12
mm
  Baseline to 3 months BIC (Mesial measurement) | -0.04 (0.08) | 0.02 (0.05)
  3 to 12 months BIC (Mesial) | 0.05 (0.10) | 0.04 (0.10)
  Baseline to 12 months BIC (Mesial) | 0.00 (0.13) | 0.06 (0.12)
  Baseline to 3 months BIC (Distal Measurement) | -0.02 (0.13) | -0.04 (0.12)
  3 to 12 months BIC (distal) | -0.07 (0.12) | 0.05 (0.08)
  Baseline to 12 months BIC (distal) | -0.08 (0.15) | 0.01 (0.12)

ADVERSE EVENTS:
Time Frame: Research related adverse events were collected throughout the study period, up to 1 year.
Arm/Group | Type 1 Implant and Thick Biotype | Type 1 Implant and Thin Biotype
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT02154581/Prot_SAP_000.pdf